CLINICAL TRIAL: NCT02013401
Title: Transmission of Discrimination-Related Stress Reactivity and Reduction From Mother to Infant
Brief Title: Transmission of Mother-Infant Stress Communication
Acronym: MIBLS
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Sponsor
Other Study IDs: 2013173
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Stress
Keywords: mother-infant dyadic regulation; stress; psychophysiology; emotion regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The central aim of this study is to assess mother-infant communication via behavioral, physiological, and affective indices under conditions where distal stressors may not be directly detectable by the infant.

DETAILED DESCRIPTION:
This investigation examines a distal maternal stressor on the quality of interaction in mother-infant dyadic communication. Assessments include behavioral, physiological, and affective indices under conditions where distal stressors may not be directly detectable by the infant. The present research examines mother-infant interactions to test the hypothesis of whether maternal stress may be transduced to their infants via multiple pathways. The secondary aim is to explore effective emotion regulation strategies for the mother as potential buffers to stress and additionally reducing early life stress effects on the infant's regulatory development.

While the emotion regulation literature posits that reappraisal may be associated with decreased in physiological and psychological stress, this type of regulation strategy may be ineffective when interfacing with discrimination. The regulation strategy needs to be titrated to the stressor in order to be effective. These findings will have notable social, clinical, and psychological significance,

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* No presence of heart murmur or wear a pacemaker
* No medication for hypertensive or cardiovascular disease
* Not using beta blockers

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of women (ages 18-40) with infants ages 4-9 months
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07-14 (Actual); Study Completion 2016-07-14 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol | One lab appointment for approximately 80 minutes.
  Salivary cortisol is a measure that indicates hypothalamus-pituitary-adrenal axis activity. The study obtains 4 assessments with 20 minutes between each assessment. Participants chew on a cotton role for 2-minutes which is placed in a cortisol salivette tube (Sarstedt)

SECONDARY OUTCOMES:
Salivary Amylase | One lab appointment for approximately 80 minutes.
  Salivary amylase is an indicator of sympathetic nervous system activity. The same salivary salivette is used to later extract the amylase.

OTHER OUTCOMES:
Mother-infant observations | One lab appointment for approximately 80 minutes.
  At four assessment occasions during the one time visit, the mother and infant are observed for a free 2-minute period. Observations include global affect, and (present or not) vocalizations, infant fussiness, and motor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kymberlee O'Brien, PhD, Principal Investigator — Postdoctoral Research Fellow; Celia L Moore, PhD, Study Director — Director of DSRC and Horizon Center; Edward Tronick, PhD, Study Director — Director Child Development Unit
Locations (2):
- United States (2):
  - University of Mass. Boston, Boston, Massachusetts
  - University of Massachusetts, Boston, Child Development Unit, Boston, Massachusetts